CLINICAL TRIAL: NCT03323151
Title: A Phase I/II Study of Ixazomib and Ibrutinib in Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: A Study of Ixazomib and Ibrutinib in Relapsed/Refractory Mantle Cell Lymphoma
Acronym: PrE0404
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0404; X16077 (Other: Takeda)
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Mantle-Cell Lymphoma
Keywords: Relapsed Mantle-Cell Lymphoma; Refractory Mantle-Cell Lymphoma; Ixazomib; Ibrutinib; Proteasome Inhibitor; Bruton's Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ixazomib; ibrutinib

STUDY DESIGN:
Intervention Model Description: Phase I: Standard 3+3 design with the primary objective of determining the maximum tolerate dose (MTD)/recommended phase 2 dose (RP2D) of this combination in MCL. Both ibrutinib-pretreated and ibrutinib-naïve patients will be enrolled.
  Phase II: Dose Level 2 is the RP2D. Patients will be enrolled to two cohorts, based on prior ibrutinib treatment: BTK-naïve and BTK-pretreated (BTK pretreated closed 8/7/2020).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I: Ixazomib & Ibrutinib (Experimental): Ixazomib and Ibrutinib will be given by mouth until progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Ibrutinib
- Phase II: Ixazomib & BTK-Naive (Experimental): Patients who are BTK-Naive will receive Ixazomib and Ibrutinib by mouth until progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Ibrutinib
- Phase II: Ixazomib & BTK Pre-Treated (Closed 8/7/2020) (Experimental): Patients previously treated with a BTK will receive Ixazomib and Ibrutinib by mouth until progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib 3 mg by mouth on days 1, 8 and 15 by mouth days 1-28 of a 28 day cycle. Dose may be escalated (Ixazomib 4 mg) dependent on dose-limiting toxicities. Note: Ixazomib dose will not be de-escalated but remain at 3 mg.
  Other Names: Ninlaro
  Arms: Phase I: Ixazomib & Ibrutinib
Drug: Ixazomib — Ixazomib 4 mg by mouth on days 1, 8 and 15 of a 28 day cycle until progression or unacceptable toxicity.
  Other Names: Ninlaro
  Arms: Phase II: Ixazomib & BTK Pre-Treated (Closed 8/7/2020); Phase II: Ixazomib & BTK-Naive
Drug: Ibrutinib — Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle. Dose may be de-escalated (Ibrutinib 420 mg) or escalated (Ibrutinib 560 mg) dependent on dose-limiting toxicities.
  Other Names: Imbruvica
  Arms: Phase I: Ixazomib & Ibrutinib
Drug: Ibrutinib — Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle until progression or unacceptable toxicity.
  Other Names: Imbruvica
  Arms: Phase II: Ixazomib & BTK Pre-Treated (Closed 8/7/2020); Phase II: Ixazomib & BTK-Naive

SUMMARY:
Patients with mantle cell lymphoma (MCL) that has relapsed (come back) or refractory (progressed on treatment) will receive ixazomib and ibrutinib.

Ibrutinib has been approved by the Food and Drug Administration (FDA) as treatment for patients with mantle cell lymphoma who have received at least one prior therapy.

Ixazomib is in a class of medications called proteasome inhibitors. Cancer cells depend on proteasome to provide this protein metabolism (turnover) function to regulate their growth and survival. Ixazomib disrupts a cancer cells' ability to survive by blocking the proteasome and disrupting protein metabolism. This may help to slow down the growth of cancer or may cause cancer cells to die.

The purpose of this study is to see whether the addition of ixazomib to ibrutinib chemotherapy is effective in treating people who have relapsed or refractory MCL and to examine the side effects associated with ixazomib in combination with ibrutinib.

DETAILED DESCRIPTION:
MCL is a rare subtype of non-Hodgkin lymphoma that is considered incurable with conventional therapy. For relapsed patients, Ibrutinib, lenalidomide, and bortezomib are all approved by the FDA but are not curative. Novel approaches are required to improve outcomes for patients with relapsed/refractory MCL.

This is an open-label study that will be done in 2 phases. Phase I will test different doses of ixazomib and ibrutinib to determine the maximum safe and tolerated dose. In Phase I, patients who have already received ibrutinib, may participate if they meet certain criteria (i.e., have not received ibrutinib for at least 3 months).

Phase II will find out the effects, good and/or bad, of ixazomib in combination with ibrutinib. In Phase II, patients will be separated into 2 groups, patients who have never received a Bruton's Tyrosine Kinase (BTK) inhibitor and patients who have received a BTK inhibitor. This study is designed to examine the effectiveness of this drug in treating patients with MCL.

Patients will be treated until progression or unacceptable toxicity.

Tumor assessments will be performed approximately every 3 months for the first year of treatment, then every 6 months until progression.

Mandatory bone marrow and tumor tissue samples (i.e., obtained during a previous procedure or biopsy) are required at baseline. Mandatory research blood samples will also be collected.

ELIGIBILITY:
* Relapsed or refractory, pathologically proven mantle cell lymphoma. Must have a current or prior tissue sample that is IHC positive for cyclin D 1 or that is positive by FISH or cytogenetics for t(11;14).
* Must have been refractory to and/or relapsed/progressed after at least 1 prior therapy.
* Prior autologous or allogeneic transplant are allowed. Patients may not have active grade II-IV acute graft-versus-host disease (GVHD) or moderate/severe chronic GVHD by NIH criteria and may not require immunosuppressive medications and/or corticosteroids for the management of acute or chronic GVHD.
* Phase I: Prior proteasome inhibitor and/or Bruton's tyrosine kinase (BTK) inhibitors are allowed but patients may not have been exposed to the combination of proteasome inhibitor and BTK inhibitor. Patients who have progressed on ibrutinib that are felt to be at high risk for rapid progression on this study shall not be eligible for the phase I portion of the study. NOTE: Ibrutinib pre-treated patients must meet all eligibility criteria AND must have discontinued prior ibrutinib at least 3 months prior to starting study therapy. PHASE I COMPLETED NOVEMBER 25, 2019.
* Phase II: Prior proteasome inhibitors allowed. (Please note prior to Version 3.0 of the protocol prior proteasome inhibitor and/or Bruton's tyrosine kinase inhibitors were allowed but patients could not have been exposed to the combination of proteasome inhibitor and BTK inhibitor).
* Age ≥ 18 years.
* Eastern Oncology Oncology Group (ECOG) performance status of 0-2.
* Ability to understand and willingness to sign Institutional Review Board (IRB)-approved informed consent.
* Willing to provide archived tumor tissue, bone marrow (if sufficient bone marrow and tumor tissue are available) and blood samples for research.
* Adequate organ function as measured by the following criteria

  * Absolute Neutrophil Count (ANC) ≥ 750/mm³
  * Platelets ˃50,000/mm³
  * Serum Creatinine ≤ 2x Upper Limit Normal (ULN)
  * ALT and AST ≤ 3x ULN
  * Total Bilirubin ≤ 1.5x ULN
* Patients must not have received systemic treatment for MCL for at least 14 days prior to enrollment, except for steroids which may be used to manage acute symptoms related to disease up to 48 hours prior to starting study therapy. Radiation therapy must be concluded at least 14 days prior to enrollment.
* Women must not be pregnant or breastfeeding since we do not know the effects of ixazomib and ibrutinib on the fetus or breastfeeding child. All sexually active females of childbearing potential must have a blood test to rule out pregnancy within 2 weeks prior to registration.
* Sexually active women of child-bearing potential with a non-sterilized male partner and sexually active men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 3 months following last dose of study drugs.
* Patients must have resolved all prior non-hematologic toxicities assessed as related to prior therapy to ≤ grade 1.
* Patients must have measurable disease (i.e., ≥ 1.5 cm in largest diameter) by conventional imaging modalities. Patients with extranodal involvement as the only measurable site of disease must have a largest diameter ≥ 1.0 cm and must be attributable to active lymphoma in the opinion of the investigator.
* Patients may not have current/active Central Nervous System (CNS) involvement with mantle cell lymphoma (patients with prior CNS involvement are eligible as long as they have had no evidence of active CNS disease for at least 6 months).
* Patients may not have another malignancy that could interfere with the evaluation of safety or efficacy of this combination. Patients with a prior malignancy will be allowed without study chair approval in the following circumstances:

  * Not currently active and diagnosed at least 3 years prior to the date of enrollment.
  * Non-invasive diseases such as low risk cervical cancer or any cancer in situ
  * Localized disease in which chemotherapy would not be indicated (such as Stage I colon, lung, prostate or breast cancer). Patients with other malignancies not meeting these criteria must be discussed with PrECOG prior to enrollment.
* Patients requiring long-term anticoagulation must be managed on an anticoagulant besides warfarin. Patients who require warfarin are not eligible.
* Patients with a clinically significant bleeding episode as judged by the investigator within 3 months of registration are not eligible, except patients who suffer bleeding due to trauma.
* Patients may not have had major surgery within 14 days, or minor surgery within 3 days, before registration.
* Patients may not have any active infection requiring oral or intravenous antimicrobial therapy at the time of therapy initiation. Patients with a recent self-limited infection that has clinically resolved may complete a prescribed course of antimicrobial therapy after study initiation as long as they are asymptomatic with no clinical evidence of infection for at least 7 days prior to treatment. Patients with a recent serious (grade ≥ 3) infection requiring hospitalization must have completed all antimicrobial therapy within 14 days of therapy initiation.
* Patients may not have evidence of uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure (New York Heart Association (NYHA) class III or higher, unstable angina, or myocardial infarction within the past 6 months. Patients with a history of any significant cardiovascular disease that has been controlled for at least 14 days before registration are allowed (except for patients who have had a myocardial infarction within 6 months).
* No systemic treatment, within 14 days before the first dose of ibrutinib with moderate or strong inhibitors of CYP3A (Strong Inhibitors: ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, and telithromycin; Moderate Inhibitors: fluconazole, darunavir, erythromycin, diltiazem, atazanavir, aprepitant, amprenavir, fosamprenavir, crizotinib, imatinib, verapamil, ciprofloxacin, grapefruit juice products, and Seville oranges) or strong CYP3A inducers for ibrutinib and ixazomib (carbamazepine, rifampin, phenytoin, St. John's wort).
* Patients with ongoing or active systemic infection, active hepatitis B or C virus infection, or known Human Immunodeficiency Virus (HIV) positive are not eligible. Testing is not required in absence of clinical suspicion.
* Patients with a history of hepatitis B or C must have a negative peripheral blood Polymerase Chain Reaction (PCR) and may not be positive for Hepatitis B surface antigen. Patients with cirrhosis or other evidence of liver damage due to Hepatitis B or C are not eligible.
* Patients with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of the treatment according to the protocol are not eligible.
* Patients with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent are not eligible.
* Patients with known gastrointestinal (GI) disease or prior GI procedure that could interfere with the oral absorption or tolerance of ixazomib or ibrutinib including difficulty swallowing are not eligible.
* Patients with ≥ Grade 2 peripheral neuropathy, or Grade 1 peripheral neuropathy with pain on clinical examination during the screening period are not eligible.
* Patients may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial throughout the duration of this study.
* As ibrutinib will not be provided by the study, the patient must be able to obtain ibrutinib through other means (i.e., commercially or through patient assistance programs). This must be confirmed prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon B Cohen, MD, Study Chair — Emory University - Winship Cancer Institute
Locations (14):
- United States (14):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Carle Cancer Center, Urbana, Illinois
  - University of Kansas, Overland Park, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU, New York, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Ixazomib & Ibrutinib (Dose Level 1): Ixazomib and Ibrutinib will be given by mouth until progression or unacceptable toxicity.
  Ixazomib: Ixazomib 3 mg by mouth on days 1, 8 and 15 by mouth days 1-28 of a 28 day cycle. Dose may be escalated (Ixazomib 4 mg) dependent on dose-limiting toxicities. Note: Ixazomib dose will not be de-escalated but remain at 3 mg.
  Ibrutinib: Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle. Dose may be de-escalated (Ibrutinib 420 mg) or escalated (Ibrutinib 560 mg) dependent on dose-limiting toxicities.
- Phase I: Ixazomib & Ibrutinib (Dose Level 2): Ixazomib and Ibrutinib will be given by mouth until progression or unacceptable toxicity.
  Ixazomib: Ixazomib 4 mg by mouth on days 1, 8 and 15 by mouth days 1-28 of a 28 day cycle.
  Ibrutinib: Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle. Dose may be de-escalated (Ibrutinib 420 mg) or escalated (Ibrutinib 560 mg) dependent on dose-limiting toxicities.
- Phase II: Ixazomib & BTK Pre-Treated: Patients previously treated with a BTK will receive Ixazomib and Ibrutinib by mouth until progression or unacceptable toxicity.
  Ixazomib: Ixazomib 4 mg by mouth on days 1, 8 and 15 of a 28 day cycle until progression or unacceptable toxicity.
  Ibrutinib: Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle until progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Started | 3 | 9 | 4 | 27
Completed | 3 | 9 | 4 | 27
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with mantle cell lymphoma (MCL) that has relapsed (come back) or refractory (progressed on treatment) will receive ixazomib and ibrutinib.
  Ibrutinib has been approved by the Food and Drug Administration (FDA) as treatment for patients with mantle cell lymphoma who have received at least one prior therapy.
  Ixazomib is in a class of medications called proteasome inhibitors. It may help to slow down the growth of cancer or may cause cancer cells to die.
Groups:
- Phase I: Ixazomib & Ibrutinib (Dose Level 1); Phase I: Ixazomib & Ibrutinib (Dose Level 2): Ixazomib and Ibrutinib will be given by mouth until progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive | Total
Number analyzed (Participants) | 3 | 9 | 4 | 27 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 6 | 9
  >=65 years | 2 | 8 | 3 | 21 | 34
Age, Continuous [Median (Full Range); unit: years] | 67 [52 to 73] | 73 [63 to 84] | 74 [58 to 77] | 70 [53 to 80] | 70 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 8 | 11
  Male | 2 | 7 | 4 | 19 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 4 | 27 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 7 | 4 | 25 | 39
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 4 | 27 | 43
Ann Arbor Stage [Count of Participants; unit: Participants] — Pathological staging of lymphoma disease where stage I describes involvement of a single nodal region or organ, stage II as involvement of two or more regions on the same side of the diaphragm, stage III as involvement of nodal regions on both sides of the diaphragm, and stage IV as diffuse extralymphatic involvement. Prognosis is worse with increasing disease stage.
  Participants
    Stage IE | 0 | 0 | 0 | 1 | 1
    Stage II | 0 | 2 | 0 | 2 | 4
    Stage III | 1 | 1 | 0 | 1 | 3
    Stage IV | 2 | 6 | 4 | 23 | 35
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). A score of 0 indicates fully active, 1 indicates restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2 indicates ambulatory and capable of all selfcare but unable to carry out any work activities, 3 indicates capable of only limited selfcare, and 4 indicates completely disabled.
  Participants
    0 | 1 | 4 | 3 | 19 | 27
    1 | 2 | 4 | 1 | 8 | 15
    2 | 0 | 1 | 0 | 0 | 1
Number of Prior Lines of Treatment [Count of Participants; unit: Participants] — This describes the number of lines of systemic treatment patients received to treat their Mantle Cell Lymphoma disease before enrolling to this study.
  Participants
    1 | 1 | 7 | 2 | 18 | 28
    2 | 1 | 1 | 1 | 5 | 8
    3 | 0 | 1 | 1 | 4 | 6
    4 | 1 | 0 | 0 | 0 | 1
MCL International Prognostic Index-c (MIPI-c) Category [Count of Participants; unit: Participants] — MCL International Prognostic Index (MIPI) is a commonly used risk stratification score that classifies patients with MCL into low-, intermediate-, and high-risk groups for overall survival. Prognosis is worst in the high-risk category.
  The MIPI-c allows to predict prognosis using clinical factors (MIPI) and the Ki-67 index. It classifies patients into these four groups: low-risk, low-intermediate-risk, high-intermediate-risk, and high-risk MCL.
  Participants
    Low | 0 | 0 | 1 | 4 | 5
    Low/Intermediate | 1 | 1 | 1 | 5 | 8
    High/intermediate and High | 2 | 5 | 2 | 18 | 27
    Indeterminate | 0 | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Dose Limiting Toxicities (DLT) Rate
Description: To determine the maximum tolerable dose (MTD) of ixazomib (mg) in combination with ibrutinib (mg) in patients with relapsed/refractory mantle cell lymphoma (MCL) using DLT endpoint.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2)
Number analyzed (Participants) | 3 | 9
Participants
  Dose Limiting Toxicity = No | 3 | 5
  Dose Limiting Toxicity = Yes | 0 | 1
  Unevaluable for Dose Limiting Toxicity | 0 | 3

2. Primary Outcome: Phase II: Complete Response Rate
Description: CR rate will be the defined as the percentage of patients achieving CR as confirmed by bone marrow biopsy within the first 12 months of initiating treatment. Response to treatment was assessed using the Lugano classification criteria. Patients completed a PET/CT at the time of study enrollment and were restaged at cycles 3, 6, 9, and 12, and then every 6 months while on study therapy.
  All patients with suspected CR who had bone marrow involvement at screening underwent a bone marrow biopsy to confirm response.
Time Frame: 12 months
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Number analyzed (Participants) | 4 | 27
Participants
  Complete Response | 0 | 11
  Partial Response | 2 | 10
  Stable Disease | 1 | 0
  Progressive Disease | 1 | 6
  Unevaluable | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Number of patients with abnormal laboratory values and/or adverse events (defined as a new untoward medical occurrence or worsening of a pre-existing medical condition) related to study treatment. Grades refer to the severity of the adverse event, where grade 1 through 5 signifies mild, moderate, severe, life-threatening, and death respectively.
Time Frame: Phase I: 12 months; Phase II: 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Ixazomib & BTK Pre-Treated: Patients previously treated with a BTK will receive Ixazomib and Ibrutinib by mouth until progression or unacceptable toxicity.
  Ixazomib: Ixazomib 4 mg by mouth on days 1, 8 and 15 of a 28 day cycle until progression or unacceptable toxicity.
  Ibrutinib: Ibrutinib 560 mg by mouth days 1-28 of a 28 day cycle until progression or unacceptable toxicity.
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Number analyzed (Participants) | 3 | 9 | 4 | 27
Participants
  Grade 1 | 0 | 0 | 0 | 1
  Grade 2 | 0 | 1 | 1 | 6
  Grade 3 | 3 | 7 | 3 | 18
  Grade 4 | 0 | 1 | 0 | 1
  Grade 5 | 0 | 0 | 0 | 1

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR assessed in accordance with Lugano classification
Time Frame: Phase I: 12 months; Phase II: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Number analyzed (Participants) | 3 | 9 | 4 | 27
Participants
  Complete (CR) or Partial Response (PR) | 2 | 6 | 2 | 21
  Non-CR/-PR | 1 | 3 | 2 | 6

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS assessed in accordance with Lugano classification
Time Frame: Phase I & II: 48 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Number analyzed (Participants) | 3 | 9 | 4 | 27
Months | 17.12 [2.56 to 36.44] | 27.43 [5.78 to 29.17] | 14.16 [2.14 to 14.16] | 29.83 [8.28 to 35.12]

6. Secondary Outcome: Overall Survival (OS)
Description: OS assessed during clinic visit or by reaching out to patients to confirm vital status.
Time Frame: Phase I & II: 48 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
Number analyzed (Participants) | 3 | 9 | 4 | 27
Months | 27.01 [20.01 to 51.15] | 47.74 [25.17 to 47.74] | 29.17 [14.16 to 37.06] | 35.68 [29.83 to 35.68]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected after each treatment cycle and for 30 days beyond treatment for up to 60 months.
Description: All serious adverse events and all-cause mortality, regardless of treatment attribution, are reported
Arm/Group | Phase I: Ixazomib & Ibrutinib (Dose Level 1) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) | Phase II: Ixazomib & BTK Pre-Treated | Phase II: Ixazomib & BTK-Naive
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/9 | 1/4 | 5/27
Serious Adverse Events (participants affected / at risk) | 2/3 | 7/9 | 1/4 | 10/27
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 4/4 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Ixazomib & Ibrutinib (Dose Level 1) (N=3) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) (N=9) | Phase II: Ixazomib & BTK Pre-Treated (N=4) | Phase II: Ixazomib & BTK-Naive (N=27)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Ixazomib & Ibrutinib (Dose Level 1) (N=3) | Phase I: Ixazomib & Ibrutinib (Dose Level 2) (N=9) | Phase II: Ixazomib & BTK Pre-Treated (N=4) | Phase II: Ixazomib & BTK-Naive (N=27)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2 | 15
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 9
Asthenia (General disorders) | 0 | 1 | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 8
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5
Fatigue (General disorders) | 1 | 4 | 3 | 16
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 1 | 0 | 0 | 7
Hypertension (Vascular disorders) | 1 | 1 | 1 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 15
Neutrophil Count Decreased (Investigations) | 1 | 2 | 0 | 4
Oedema Peripheral (General disorders) | 0 | 2 | 0 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 7
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 2 | 0 | 4
Platelet Count Decreased (Investigations) | 1 | 2 | 2 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 6
Syncope (Nervous system disorders) | 0 | 0 | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 2
Chills (General disorders) | 1 | 1 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 5
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03323151/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT03323151/SAP_002.pdf